CLINICAL TRIAL: NCT01773577
Title: The Effect of Interoperable Health IT on Efficiency in Ambulatory Practices
Acronym: HEAL5
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: State University of New York at Buffalo (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: HITEC/HEAL5
Record Dates: First submitted 2011-08-02; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2012-03

CONDITIONS: Operations Research Workflow
Keywords: EHR; VHR; Electronic Health Record

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physician Pract. Employee and Off. Staff: The office staff and providers and physician practices enrolled in the RHIO

SUMMARY:
Goal: To evaluate the effects of Interoperable Health IT on provider work flow and work practices in the ambulatory care setting.

Interoperable health IT can produce a reduction of barriers in the exchange of health information that can allow for more efficient, timely, and a higher quality of patient care. This study seeks to evaluate the effects of the implementation of interoperable health IT on the work flow of medical providers in the care environments in which they are implemented.

DETAILED DESCRIPTION:
Interoperable health IT allows for the reduction of barriers in the exchange of health information. Substantial work flow efficiencies and cost reductions may be realized by reducing these barriers, and integrating information exchange among different providers and healthcare systems. Some of the avenues in which these efficiencies and cost reductions are likely to be achieved are through easier access to test results, reduction in medication errors, quality monitoring and improvement methodologies, and increased consumer choice. In recognition of the potential for these improvements, New York State has provided funding to regional entities (Regional Health Information Organizations-RHIO'S) whose role is to assist practice providers in the development, implementation, and integration of these interoperable IT systems. New York State has also provided funding to evaluate the technology implementations facilitated by the RHIOs. The investigators will be working with health care providers that have been assisted by the Greater Rochester RHIO.

Depending on the unique characteristics of the hardware and software that is developed and implemented, there may be variations in operational flow that effect efficiency in the ambulatory care setting. The goal of our study is to measure and evaluate the effects of interoperable IT systems in the work flow practices of providers that have implemented them in the ambulatory care setting.

ELIGIBILITY:
Inclusion Criteria:

* Our population will include all of the providers and office workers within the ambulatory care settings that have implemented the interoperable IT programs, and are required to utilize the systems for their daily job functions. Our research population will not include patients, as the participants of our study are the health care workers.

Exclusion Criteria:

* Our population will be "all inclusive" of all office staff and providers that are required to utilize the systems in place in order to perform their day-to-day functions. There will be no exclusions except for those under 18 years of age, and non English speakers (neither of which are expected to be in the eligible population).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care and primary care specialty practices participating in EHR/VHR in the Rochester Regional Health Information Organization
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in workflow pattern | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Crane, MD, MBA, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States